CLINICAL TRIAL: NCT01439035
Title: Pilot Study to Evaluate Use of Optical Frequency Domain Imaging (OFDI) for Duodenal Imaging in Celiac Disease in Children, Adolescents and Young Adults
Brief Title: Evaluate the Use of Optical Frequency Domain Imaging (OFDI) for Celiac Disease in Children, Adolescents and Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Guillermo Tearney, Professor of Pathology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2009-P-000938
Record Dates: First submitted 2011-09-20; First posted 2011-09-22 (Estimated); Results first posted 2018-09-26 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Celiac Disease
Keywords: Celiac Disease; Duodenal; OCT; Imaging
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MGH OFDI imaging (Experimental): OFDI imaging
  Interventions: Device: MGH OFDI Imaging

INTERVENTIONS:
Device: MGH OFDI Imaging — Imaging of Duodenum with OFDI system

SUMMARY:
The goal of this research is to conduct a pilot clinical study to image Celiac disease characteristic mucosal lesions and compare Optical Frequency Domain Imaging (OFDI) images to histologic evaluation in children, adolescents and young adults with suspected Celiac disease.

DETAILED DESCRIPTION:
The Optical Frequency Domain Imaging(OFDI) catheter will be used in conjunction with a standard pediatric endoscope. The endoscopist will introduce the OFDI imaging catheter through the biopsy channel of the endoscope already in place. The catheter will be passed into the view of the endoscope so that the tip of the catheter can be directly visualized throughout the procedure. The catheter will be placed adjacent to the bowel wall in the vicinity of the target locations. Once the OFDI probe is in place, OFDI imaging will start and data will be continuously collected during helical pullback scanning of the inner catheter drive shaft over a predetermined length of approximately 3 cm.

It is expected that the total experimental procedure including the insertion of the OFDI catheter, OFDI imaging, and removal of the catheter will add approximately 10 minutes to the total length of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age 7 years and above undergoing upper endoscopy for evaluation of celiac disease
* Clinical history, physical findings, family history, or serologic evaluation suggestive of celiac disease
* Parents/guardian available to sign informed consent

Exclusion Criteria:

* Patients with a history of hemostasis disorders
* Use of Nonsteroidal anti-inflammatory drugs(NSAIDS) within ten days preceding initiation of the study
* Use of any oral anticoagulation medication within one month preceding initiation of the study
* Any known blood coagulation disorder

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-08; Primary Completion 2010-02-04 (Actual); Study Completion 2011-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Tearney, MD PhD, Principal Investigator — Massachusetts General Hospital; Aubrey Katz, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MGH OFDI Imaging
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | MGH OFDI Imaging
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants] — Six subjects completed this study
  Participants
    <=18 years | 4
    Between 18 and 65 years | 2
    >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.3 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Changes of Villous Architecture Undergoing OFDI Imaging
Description: OFDI images analyzed and compared to standard of care biopsies to identify celiac disease caracteristic mucosal lesions.
  In this pilot study, we demonstrated the feasibility of using OFDI for visualizing changes of villous architecture in CD patients in vivo
Time Frame: during imaging session
Population: Subjects 7 or over 7 years old with Celiac Disease
Measure: Count of Participants; unit: Participants
Groups:
- Compare OFDI Images to Histologic: compare OFDI images to histologic evaluation in children, adolescents and young adults with suspected Celiac disease
Arm/Group | Compare OFDI Images to Histologic
Number analyzed (Participants) | 6
Participants | 6

ADVERSE EVENTS:
Time Frame: The duration of the imaging procedure
Description: No adverse evens has been reported
Arm/Group | MGH OFDI Imaging
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No